# STATISTICAL ANALYSIS PLAN STUDY KCE-16012

THE USE OF A SILICONE ADHESIVE MULTILAYER FOAM DRESSING AS AN ADJUVANT PROPHYLACTIC THERAPY FOR PRESSURE ULCER PREVENTION: A MULTICENTRE RANDOMISED OPEN LABEL PARALLEL GROUP MEDICAL DEVICE TRIAL IN HOSPITALISED PATIENTS AT RISK OF PRESSURE ULCER DEVELOPMENT

This document is based on the statistical section of the protocol.

Any deviations from this plan will be described in the final clinical study report.

Version FINAL Date 05 11 2019

#### Authors:

France Vrijens (KCE, statistician)
Isabelle Savoye (KCE, data manager)

#### Reviewed by

Dimitri Beeckman (U Gent, Chief Investigator KCE 16012 study) Frank Hulstaert (KCE, MD, Senior Researcher Trials) Jilly Harrison (KCE, Researcher Trials)

ClinicalTrials.gov NCT03442777

# ■ TABLE OF CONTENTS

| 1 | INTRO | DDUCTION | 3 |
|-----|-------|--------------------------------------------|----|
| 2 | BACK | (GROUND | 3 |
| 3 | TRIAL | L OBJECTIVES AND DESIGN | 3 |
| 3.1 | STUD | Y DESIGN | 3 |
| 3.2 | | NT ELIGIBILITY CRITERIA | |
| | 3.2.1 | Inclusion criteria | 4 |
| | 3.2.2 | Exclusion criteria | 5 |
| 3.3 | SAMP | LE SIZE CALCULATION | 5 |
| 4 | DATA | NBASE | 6 |
| 5 | ANAL | .YSES | 6 |
| 5.1 | ENDP | OINTS | 6 |
| 5.2 | ANALY | YSIS POPULATIONS (ITT AND PP) | 7 |
| 5.3 | STATI | STICAL ANALYSES | 8 |
| | 5.3.1 | General considerations | 8 |
| | 5.3.2 | Demographics and baseline characteristics. | 8 |
| | 5.3.3 | Efficacy evaluation | |
| | 5.3.4 | Health economics evaluation | 10 |
| | 5.3.5 | Safety evaluation | 10 |
| 6 | CLINI | CAL STUDY REPORT | 10 |
| | APPE | NDICES | 10 |

# 1 INTRODUCTION

This document gives a detailed statistical analysis plan for the Pressure Ulcer Prevention study (KCE-16012), and should be read in conjunction with the current protocol.

# 2 BACKGROUND

A pressure ulcer is defined as a localized injury to the skin and/or underlying tissue usually over a bony prominence, as a result of pressure, or pressure in combination with shear (National Pressure Ulcer Advisory Panel, 2014). To prevent the development of pressure ulcers, the KCE clinical practice guideline recommends to reduce both the amount and the duration of pressure and shear (Beeckman, Matheï, Van Lancker, Van Houdt, Vanwalleghem et al., 2013). Currently, interest is growing in the application of multilayer foam dressings (initially being used for wound treatment) as an adjuvant prophylactic therapy for pressure ulcer prevention. The clinical effectiveness of a multilayer foam dressing as a preventative intervention for pressure ulcers has been summarized in three systematic reviews (Clark et al., 2014; Davies, 2016; Moore & Webster, 2013). The three reviews concluded at the lack of a large randomized study to ascertain the most appropriate patient populations, and anatomical locations for the use of multilayer foam dressings as a preventative intervention for pressure ulcers. The smaller trials on the prevention of pressure ulcers, providing some proof of concept, were limited to the ICU setting. The study aims to confirm the effectiveness of such intervention in ICU and non-ICU settings.

# 3 TRIAL OBJECTIVES AND DESIGN

The Pressure Ulcer Prevention trial is a multicentre, randomised, open-label trial with the following objective:

#### **Primary objective**

The objective of this study is to determine if silicone adhesive multilayer foam dressings applied to the sacrum, heels and greater trochanter in addition to standard prevention reduce pressure ulcer incidence category II, III, IV, Unstageable and Deep Tissue Injury (DTI) compared to standard pressure ulcer prevention alone, in at risk hospitalised patients. In particular, this trial extends previous trial results obtained in ICU setting.

No secondary objectives have been formulated for this trial.

#### 3.1 Study design

This is a randomised, open label, parallel group, superiority, multicentre post-marketing study. There are two intervention groups (Allevyn® and Mepilex®) and one control group (standard of care). Patients have been randomised in a 1:1:1 ratio to the Allevyn®, Mepilex® and control group and stratified by hospital and the type of ward (ICU vs non- ICU). The duration of the intervention period is maximum 14 days (see Figure 1). There is no follow-up after the end of the intervention period.



Figure 1: Study design.

#### 3.2 Patient Eligibility criteria

#### 3.2.1 Inclusion criteria

Following inclusion criteria will be applied:

- At risk for pressure ulcer development based on Braden risk assessment (Braden score ≤17).
- 2. Admitted to hospital within the previous 48 hours.

Note: Not more than 25% of patients per site should be recruited at ICU wards.

- Skin at sacrum is assessable and there is no clinically relevant incontinence- associated dermatitis (IAD) or another skin condition that would be a contra-indication for the application of the devices under study, and there is no pressure ulcer category II or worse present.
  - \*clinically relevant IAD is defined as any of the 4 categories described in the publication <a href="http://users.ugent.be/~dibeeckm/globiadnl/nlv1.0.pdf">http://users.ugent.be/~dibeeckm/globiadnl/nlv1.0.pdf</a>
- 4. for at least 3 of the following 4 skin sites (heel left, heel right, greater trochanter left, greater trochanter right) one of the following two conditions should apply:
  - A study dressing can be applied as prevention of a pressure ulcer category II or worse at that skin site (there is no contra-indication)

OR

- o There is already a pressure ulcer category II or worse at that skin site.
- 5. Written informed consent by the patient or his/her legal representative.

#### 3.2.2 Exclusion criteria

Following exclusion criteria will be applied:

- 1. Aged < 18 years.
- 2. The length of stay counting from first day of admission in one or (if the patient is transferred to another ward) more participating wards is < 7 days.
- 3. Both heels amputated
- 4. Previously known/documented allergy for substances used in the devices under study.
- 5. A clinical condition not allowing participation in a clinical study.
- 6. Participation in another interventional clinical trial.
- 7. Patients who exceptionally receive or are planned to receive a dressing for the prevention of pressure ulcers at sacrum, heels and trochanters based on best medical judgment and outside of the surgery setting.

#### 3.3 Sample size calculation

For all analyses, both treatment groups will be pooled into one group unless specified otherwise. The sample size calculation is based on this assumption.

The primary objective is to compare the incidence rate of occurrence of at least one new pressure ulcer category II, III, IV, Unstageable, and DTI pressure ulcer at sacrum, heels and greater trochanter in both treatment arms versus the control arm.

The primary hypothesis is that the incidence rate of new pressure ulcer category II, III, IV, Unstageable, and DTI at sacrum, heels and greater trochanter will be lower in the treatment groups compared to the standard of care group. Superiority will be concluded if the primary variable is significantly different in the treatment groups compared to the standard of care group, based on a two sided test at 5% level of significance.

The sample size calculation is based on the results of a number of randomised trials with data about pressure ulcer category II, III, IV, Unstageable, and DTI incidence.

- The pressure ulcer category II, III, IV, Unstageable, and DTI incidence rate on sacrum, greater trochanter and heels is 6% in the standard of care group (Schoonhoven et al., 2007)
- The treatment groups will have a 50% reduction in pressure ulcer incidence category II, III, IV, Unstageable, and DTI incidence on sacrum, greater trochanter and heels. (Demarré et al., 2012; Nixon et al., 2006)

In order to have 80% power to show superiority, data should be available for 1578 patients in total of which 526 are allocated to the control group and 1052 are allocated to the treatment group.



Considering approximately 5% drop a total of 1662 patients are to be randomised to ensure that sufficient patients complete the study without compromising the power of the study.

Exploratory efficacy analysis will compare the effectiveness of the two treatments: Allevyn® and Mepilex®. The null hypothesis is that there is no difference between Allevyn® and Mepilex®. The alternative hypothesis is that there is a difference between the treatment groups. The difference will be tested two- sided at 5 % level of significance.

# 4 DATABASE

The database comprises of the following 9 datasets:

#### Clinical Database

- 1. GEN (GENERAL): general datasets with all demographics and inclusion and exclusion criteria, 1 line per patient (contains all patients who consented to the study)
- 2. ASS (ASSESSMENTS): all the assessments data, 1 line per patient per day.
- 3. PHO (PHOTOS): central blinded review of the pictures (the pictures will also be transferred).
- 4. ADE (ADVERSE EVENT DEVICE): 1 line per reported case. All descriptions are in free text.
- 5. DD (DEVICE DEFICIENCY): one line per reported case.
- 6. COM (COMMENTS in e-CRF) one line per comment

#### Data Management and Monitoring Database

- 7. DCR (DATA CLARIFICATIONS REQUEST), 3 types of requests (Monitor; automatic edits checks; Data management). 1 line per DCR.
- 8. MONITORING: information on whether the page has been monitored or not on site.

#### **Audit Trail**

9. A\_TRAIL (AUDIT TRAIL): audit trial of whole eCRF. It contains all the creation of records and the changes that have been made to it, when and by whom.

The annotated e-CRF describes all variables present in the database (see appendix 1).

All datasets are in SAS format (extension .sas7bdat).

# 5 ANALYSES

# 5.1 Endpoints

The following endpoints will be analysed:

#### Clinical endpoints

- Occurrence of a new Pressure Ulcer category II or worse (i.e. a Pressure Ulcer Category II, III, IV, Unstageable, and Deep Tissue Injury) at any site during the observation period, as reported by site.
- 2. Occurrence of a new Pressure Ulcer category II or worse (ie Pressure Ulcer Category II, III, IV, Unstageable, and DTI) on sacrum, right greater trochanter, left greater trochanter, right heel, left heel during the observation period, <u>as reported by site</u>.



3. Occurrence of a new Pressure Ulcer category II or worse (i.e. a Pressure Ulcer Category II, III, IV, Unstageable, and Deep Tissue Injury) at any site and by body site, during the observation period, as confirmed by central review of pressure ulcer pictures.

For all those endpoints, a patient with a PU (cat II or above) already present at baseline for the specific site assessed will be excluded for the analysis of that specific site. For patients with a specific site not assessable at baseline, the first day where this site is assessed will be used as baseline information.

#### Health Economics endpoints

- 4. Area under the curve for utilities derived from EQ-5D-5L Quality of Life score at Day 3 and Day 14 or end of study day.
- 5. Number of dressing applied during intervention period (by body site and in total), for patients versus pressure ulcers prevented overall and by body site.

#### Safety endpoints (only for patients in the intervention group)

- 6. Occurrence of any Adverse Device Effect (ADE)
- 7. Occurrence of any Serious Adverse Device Effect (SADE)
- 8. Occurrence of any Device Deficiency (DD)

# 5.2 Analysis populations (ITT and PP)

The following analysis sets will be considered:

- 1. **Total Set**: all patients who consented to participate in the study and who did not explicitly ask to have their data excluded from the analysis.
- 2. Intent-to-treat (ITT) Population: All patients of the Total set who were randomised.
- Per Protocol (PP) Population: all patients of the ITT Population who received the study treatment according to the protocol, without any major protocol deviation impacting the primary efficacy assessment.
- 4. **Safety Population**: all patients of the ITT population who entered into the observation period and who were applied at least once dressing.

For the ITT Population patients will be considered in the treatment group as randomised (as foreseen by the attributed randomisation number). For the other analysis sets patients will be considered in the treatment group as treated.

The efficacy analyses will primarily be performed for the ITT Population and supportively for the PP Population

For the PP analyses, patients will be excluded:

- 1. If they were non-eligible for the study (if they did not meet all inclusion criteria, or they met one of the exclusion criteria )
- 2. who received the intervention of another group (not the one allocated using randomisation)
- 3. patients who were not applied any dressing during the intervention period on the specific site assessed
- 4. who discontinued the intervention for any reason before day 3 (as pressure ulcer incidence is likely highest on day 3)



#### 5.3 Statistical analyses

#### 5.3.1 General considerations

The statistical analysis will be performed using the SAS statistical package, version 9.2.

#### **Descriptive statistics**

Unless otherwise stated, summary statistics for quantitative variables will include the mean, standard deviation, minimum, 1st quartile, median, 3rd quartile, maximum, number of observations, and number of missing values. For categorical variables absolute counts (n) and percentages (%) of patients with data will be presented.

#### P-values

Unless otherwise specified, all p-values will be from two-sided test. No corrections for multiple testing will be made.

#### Missing data

Patients without any assessment of the primary endpoint after randomization will be excluded from the ITT population.

#### 5.3.2 Demographics and baseline characteristics.

A description will be given of key patient characteristics recorded at the baseline visits, for all patients and broken down by treatment group. See appendix 2 for templates of tables' results.

The following conventions will be taken take

- Age: is the age at the date of written informed consent.
- Time spent is hospital: is the time from data of hospital admission to the date of written informed consent (maximum 48 hours per protocol)
- Time since surgery: is the time from data of surgery to the date of written informed consent
- BMI will be categorized following usual international standards
- Braden Score at baseline will be categorised as mild risk (17), moderate risk (12-16), low risk (11 and lower)

#### 5.3.3 Efficacy evaluation

#### Primary efficacy variable

For the primary efficacy variable:

 Comparison of the treatment group (Allevyn® & Mepilex® pooled) versus the control group (incidence rate is frequency at which patients develop one or more such new pressure ulcers over the study period as judged on site) by means of the CMH test controlled for type of ward (ICU/Non-ICU).

Patients in study arms 1 and 2 will be pooled as the treatment group and the incidence rate of pressure ulcers category II or worse as judged on site will be compared between the treatment group and the usual care group as per randomisation scheme, by means of the CMH test controlled for type of ward (ICU/Non-ICU).



The primary endpoint of this study is the incidence rate during the study period of the patient (during maximum 14 days) of at least one new pressure ulcer category II, III, IV, Unstageable, Deep Tissue Injury (DTI) (briefly referred to as pressure ulcers category II or worse) on sacrum, heels and greater trochanter as judged on site. The primary analysis of the primary efficacy variable is a superiority analysis that compares the incidence rate in the pooled treatment groups versus the control group, on the ITT population by means of the CMH test controlled for type of ward (ICU/Non-ICU). Superiority will be concluded if the estimated impact of the treatment (Allevyn® and Mepilex® versus standard of care) is significant based on a 2 sided test at 5% significance level.

#### Subgroup analyses of primary endpoint

#### All sites

Subgroup analyses will be performed on the following variables:

- Age (<60, 60-69, 70-79, 80+)
- Gender
- Ward (ICU, non-ICU)
- Surgery (yes/no)
- BMI (categories)
- Diabetes (yes/no)
- By Braden Scale Score at baseline (17, 12-16, 11 or less), and by Braden score specific dimensions:
  - Nutrition (very poor or probably inadequate versus adequate or excellent)
  - Sensory perception (completely limited or very limited versus slightly limited or no impairment)
- Activity (bedfast or chairfast versus walks occasionally or walks frequently)
- o Mobility (completely immobile or very limited versus slightly limited or no limitations)
- Hospital

#### In addition, for the analysis of the sacrum and the trochanters

By Braden score for

Moisture (constantly moist or very moist or occasionally moist versus rarely moist)

#### In addition, for the analysis of the heels

By Braden score for

o Friction and shear (problem or potential problem *versus* no apparent problem)

These exploratory subgroup analyses will be undertaken, appropriately cautiously, to investigate any influence of the prognostic factors.

See appendix 3 for templates of tables' results on clinical endpoints.

#### Sensitivity analysis

• A sensitivity analysis will be conducted in the ITT populations based on the reviewed photographs of the PU, based on the review by the CI team.

#### **Exploratory analyses**

 Comparison (ITT and PP) of incidence rates (primary endpoint) between the experimental investigational devices (arms 1 and 2). Statistical Analysis Plan: KCE-16012

#### Exploratory efficacy variables: logistic regression

A sensitivity analysis will be done using logistic regression. The model of the logistic will have the following variables: intervention group, hospital, age, sex, type of ward and Braden score category. A comparison between the efficacy of the two treatments will be made by defining a contrast in the logistic model. A difference between the two treatments will be concluded if there is a significant difference between the two treatments based on 2 sided testing at the 5% significance level.

#### 5.3.4 Health economics evaluation

Health economic analyses will be performed on the basis of the ITT population.

Because no Belgian values for the EQ5D utilities<sup>a</sup> are currently available (this is an undergoing project at KCE), values from The Netherlands will be used (with a sensitivity analysis based on values from England).

Statistical comparisons on the impact of the intervention on the QOL will be for exploratory purposes only.

No statistical comparison will be performed on the number of dressings applied.

See appendix 4 for templates of tables' results on health economics endpoints.

#### 5.3.5 Safety evaluation

Safety analyses will be performed on the basis of the Safety Population and will be descriptive.

The description of safety findings will be provided as entered in the e-CRF (as a free text in Dutch).

No statistical comparisons will be performed on the safety endpoints.

See appendix 5 for templates of tables' results on safety endpoints.

#### 6 CLINICAL STUDY REPORT

The clinical study report will be written by the Chief Investigator. After database lock, all tables described in appendices 2 to 5 will be provided in RTF format to him.

# APPENDICES

The appendices of this SAP are in a separate document.

<sup>&</sup>lt;sup>a</sup> https://eurogol.org/eg-5d-instruments/eg-5d-5l-about/valuation-standard-value-sets/



# APPENDICES STATISTICAL ANALYSIS PLAN STUDY KCE-16012

THE USE OF A SILICONE ADHESIVE MULTILAYER FOAM DRESSING AS AN ADJUVANT PROPHYLACTIC THERAPY FOR PRESSURE ULCER PREVENTION: A MULTICENTRE RANDOMISED OPEN LABEL PARALLEL GROUP MEDICAL DEVICE TRIAL IN HOSPITALISED PATIENTS AT RISK OF PRESSURE ULCER DEVELOPMENT

This document contains the appendices of the statistical analysis plan.

Version FINAL Date 08 10 2019

#### Authors:

France Vrijens (KCE, statistician)
Isabelle Savoye (KCE, data manager)

#### Reviewed by

Dimitri Beeckman (U Gent, Chief Investigator KCE 16012 study) Frank Hulstaert (KCE, MD, Senior Researcher Trials) Jilly Harrison (KCE, Researcher Trials)



# **■ TABLE OF CONTENTS**

| APPE | NDICES | 3 |
|-------------|------------------------------------------------------|----|
| | ANNOTATED E-CRF | |
| APPENDIX 2. | TEMPLATE TABLES RESULTS (1) PATIENT INFO | 32 |
| APPENDIX 3. | TEMPLATE TABLES RESULTS (2) CLINICAL OUTCOMES | 50 |
| APPENDIX 4. | TEMPLATE TABLES RESULTS (3) HEALTH ECONOMIC OUTCOMES | 56 |
| APPENDIX 5. | TEMPLATE TABLES RESULTS (4) SAFETY OUTCOMES | 58 |

The tables templates presented in this SAP are based on the analysis of a mock database of 10 patients. The tables in the final clinical study report may look slightly different in function of the analysis of the complete database.

# ■ APPENDICES

# **APPENDIX 1. ANNOTATED E-CRF**



#### **Annotated CRF for**

THE USE OF A SILICONE ADHESIVE MULTILAYER FOAM DRESSING AS AN ADJUVANT PROPHYLACTIC THERAPY FOR PRESSURE ULCER PREVENTION: A MULTICENTRE RANDOMISED OPEN LABEL PARALLEL GROUP MEDICAL DEVICE TRIAL IN HOSPITALISED PATIENTS AT RISK OF PRESSURE ULCER DEVELOPMENT.

Protocol KCE-16012 (KCE2)

| Version | sion Date | | Status |
|---------|-----------|------------------|-------------|
| 1.0 | | 14 December 2017 | Final |
| 2.0 | | 12 February 2018 | Amendment 1 |
| 3.0 | | 23 March 2018 | Amendment 2 |

#### ANNOTATION OF ECRF DATABASE

#### Color code:

- Red = Variable name, with variable type between brackets
- Green = Format/codes attributed to variables
- Blue = Panel names / content
- Black = Additional documentation

#### Variable type:

 Ax: Refers to text variables that can capture integers (e.g. numerical variables without decimals) with x digits, and predefined text codes such as 'NA', 'ND', etc.

#### Example: A2

- Allows entering numeric values between -9 and 99
- Allows entering text codes 'NA', 'ND', etc.
- Refuses the entry of -10.
- Ax.y: Refers to text variables that can capture numeric values, with x the width of the field (including the decimal field separator '.') and y the maximum number of digits to the right of the decimal point in the numeric value, as well as predefined text codes such as 'NA', 'ND', etc.. The entry of at least one number before the decimal field separator is mandatory, the entry of the decimal field separator or of decimals is not mandatory. Information is stored as entered. When using this format for variables calculated by the system, results are always rounded to and displayed on screen with y decimals.

#### Example: A4.1

- Allows entering numeric values between -9.0 and 99.9
- Allows entering text codes 'NA', 'ND', etc.
- Accepts the entry of an integer value (values between 0 and 9999) and stores the information without adding a decimal to the value e.g. 4 is stored as '4'
- Refuses the entry of '4.12' and of '.1'.
- AFx.y: Refers to text variables that can capture numeric values, with x the width of the
  field (including the decimal field separator '.') and y the fixed number of digits to the
  right of the decimal point in the numeric value, as well as predefined text codes such as
  'NA', 'ND', etc.. The entry of the at least one number before the decimal field separator
  is mandatory, and the entry of the y decimals is mandatory.

#### Example: AF4.1

- Allows entering numeric values between -9.0 and 99.9
- Allows entering text codes 'NA', 'ND', etc.
- Refuses the entry of values with more/less than 1 decimal (e.g. 4, 4.12)

- Refuses the entry of '.1'.
- Cx: Refers to text variables of length x. Can consist of letters (lower and upper case), numbers or any combination of these. While exporting the data, special characters (ASCII characters 8, 9, 10, 11 and 13) are replaced by a space.

#### Example: C255:

- Allows entering any text string of maximum 255 characters.
- Nx: Refers to integers (e.g. numerical variables without decimals) with x digits

#### Example: N2:

- Allows entering numeric values between -9 and 99.
- Refuses the entry of text codes 'NA', 'ND', etc.
- Refuses the entry of -10.
- Nx.y: Refers to numerical variables, with x the width of the field (including the decimal field separator '.') and y the maximum number of digits to the right of the decimal point in the numeric value. The entry of at least one number before the decimal field separator is mandatory, the entry of the decimal field separator or of decimals is not mandatory. Information is stored as entered. When using this format for variables calculated by the system, results are always rounded to and displayed on screen with y decimals.

#### Example: N4.1:

- Allows entering numeric values between -9.0 and 99.9.
- Allows the entry of an integer value (values between 0 and 9999) and stores the information without adding a decimal to the value e.g. 4 is stored as '4'; Refuses the entry of '4.12' and of '.1'
- Refuses the entry of text codes 'NA', 'ND', etc..
- NFx.y: Refers to numerical variables, with x the width of the field (including the decimal field separator '.') and y the number of digits to the right of the decimal point in the numeric value. The entry of at least one number before the decimal field separator is mandatory, and the entry of the y decimals is mandatory.

#### Example: NF4.1:

- Allows entering numeric values between -9.0 and 99.9.
- Refuses the entry of Text codes 'NA', 'ND', etc.
- Refuses the entry of values with more/less than 1 decimal (e.g. 4, 4.12)
- Refuses the entry of '.1'.

#### Notes:

- For variables of type A and N:
  - If decimal parts are allowed, the point ('.') should be used as decimal field indicator. The use of a thousand field indicator is not allowed.
- · For variables of type A:
  - When entering leading zero's, these will be retained and considered when verifying whether the entry fits in the maximal width allowed for the variable.
  - Leading zero's may be entered, but are not mandatory to be entered, except if otherwise documented in the screen or edit check plan document.
- For variables of type N:
  - When entering leading zero's, these will be removed and not considered when verifying whether the entry fits in the maximal width allowed for the variable.

#### DOCUMENT HISTORY

#### Amendment 1:

- 1.7 Inclusion / Exclusion Criteria:
  - · New variable ECT7 added
  - · Text of ICT3 and ICT4 has changed
  - Changed IC1-IC5 into ICT1-ICT5 and EC1-EC7 into ECT1-ECT7
  - Changed ARM[C1] into ARM[C16]
  - · Added variables for date of randomisation and time of randomisation

#### - 1.9 Daily assessment:

- Section Study Intervention: Variables for 'Dressing type applied' changed from tickboxes to numerical fields
- Corrected the length for SUPSURFT, FREQREPT, COMPIDT

#### - 1.10 Termination:

- · 'Date of end of study intervention on ALL body sites' changed from N to A
- 1.11 Adverse Device Effects (ADE) Log:
  - Corrected the length for ADEOUTT
- 1.14 Device Deficiency (DD) Log:
  - · Corrected the length for DDNAT

#### Amendment 2:

- 1.13 Photographs Log: annotation added
- Photographs Log for Blind Review: annotation added
- 1.9: format of Day changed from [N1] into [C3]

# FLOW OF THE E-CRF SCREENS

# Creation of patient

| | Screen |
|-----|------------------|
| 1.4 | Informed Consent |

# Day 1 (Baseline)

| | Screen |
|-----|--------------------------------------|
| 1.5 | Patient Profile |
| 1.6 | Pre-Randomisation Assessment (Day 1) |
| 1.7 | Inclusion / Exclusion Criteria |
| 1.8 | Day 1 – Study Intervention |

# Day 2 until Day 14

| | Screen |
|-----|------------------|
| 1.9 | Daily Assessment |

# Log Screens

| | Screen | a |
|------|----------------------------------|---|
| 1.10 | Termination | |
| 1.11 | Adverse Device Effects (ADE) Log | 9 |
| 1.12 | Comments Log | 9 |
| 1.13 | Photograph Log | |
| 1.14 | Device Deficiency (DD) Log | |
| 1.15 | Investigator Statement | |

# Reviewer Screen

| Screen |
|----------------------------------|
| Photographs Log for Blind Review |

# 1.1. Log-on to the System

# 1.1.1. Screen

| Jser ID |
|---|
| Password |
| The second secon |
| The password to have access to this e-CRF is personal and confidential. It should not be shared with any third party. |
| □ I understand and agree with these conditions |
| LOGIN |
| Activate Account |
| If you have an activation code, you can activate your account here |
| Reset Password |

#### 1.2. Patients Overview

#### 1.2.1. Screen

| Patients | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Add ne | w patient | Searc | ch |
| Patient ID | Ward upon<br>enrollment | User who randomised | Last day<br>assessed or<br>EOS status | Status | Active | PDF | Ready for sign-off | Details |
| Y . | | | | | | | Ready | |

Annotated CRF for protocol KCE-16012 (KCE2)

1.3. Patient Summary

#### 1.4. Informed Consent

# PATIENT\_ID = SUBJID[C7]

1.4.1. Screen

| Informed Consent DCONSD[N2] DCONSM[N2] DCONSY[N | 14] ———— |
|---|---|
| Date of written informed consent: (dd) (mm) (yyyy) | , a |
| EDITCONS[N1] Trick in case the date of written informed consent needs to be of | corrected |
| 1= Ticked Corrected date of written informed consent: (dd) (mm) (y) | DCONS2D[N2] DCONS2M[N2] DCONS2Y[N4 |
| Informed consent signed by: 1 = Ticked □ Legal representative CONSREP[N1] | |
| Ward on which the patient is staying upon enrollment: | 2<br>C Non-ICU WARD[N1] WARDT[C7] |
| EDITWARD[N1] Tick in case the ward needs to be corrected 1 Ticked Corrected ward: CICU | 2<br>C Non-ICU WARD2[N1] WARD2T[C7] |
| Back | Save Save and Next |

# 1.5. Patient Profile

#### 1.5.1. Screen

| Date of birth: DDE | BD[A2] DD | BM[A2] | DDBY[N4] |
|---|---|---|---|
| Gender: 1 C Male 2 C Female S | EX[N1] SEX | XT[C6] | |
| Height: | | cm | HEIGHT[A3] |
| Weight: | | kg | WEIGHT[A5.1] |
| Body Mass Index (BMI): | | | BMI [N4.1] |
| Does the patient have diabetes? | ○ Yes | O No<br>2 | DIABETE[N1] DIABETET[C3] |

# 1.6. Pre- Randomisation Assessment (Day 1)

1.6.1. Screen

| Pre - Rando | misation As | sessment (C | ay 1) | | | | | , |
|---|---|---|---|---|---|---|---|---|
| Date (do | d) (mm) (yy | | IDD[N2] DRA | ANDM[N2] | DRANDY | [N4] | | |
| 1. Admissio | n informatio | n DADME | [N2] DADM | M[N2] DA | DMY[N4] | | | |
| Date admiss | sion to hospita | al: (de | d) (mm) (yyyy) | | Time: TAD | (hh on 24 hour o<br>MH[N2] | clock) | |
| Expected ler | ngth of stay or | n participating | wards since da | ate of admis | sion to hospi | al: 1 C Less tha | • | STAY[N1]<br>STAYT[C1 |
| Did the patie | ent have surge | ery since adm | ission? | | | 1] SURGT[ | C3] | |
| Date of | start of surge | | mm) (yyyy)<br>SURM[N2] D | 1 2<br>SURY[N4] | £ | | | |
| Type of | surgery: | 1 O Elec<br>2 O Non | SUI | RTYPE[N1 | ] SURTY | PET[C12] | | |
| Anaesth | iesia | 1 C Gen<br>2 C Loca | | RANAE[N1 | ] SURAN | AET[C7] | | |
| 2. Braden s | cale assess | ment DA | Y[N2] = 1 | REFER | O SCREE | N 1.9 | P | ANEL = ASS |
| Sensory per | ception: | Moisture: (1) | Activity: ① (1-4) | Mobility: (1-4) | Nutrition: (1-4) | Friction & she | ear <b>()</b> Brad | den score<br>(6-23) |

2=Heel right

3=Heel left 4=Greater trochanter right

5=Greater trochanter left

PANEL = ASS

| | Sacrum | Patient's right<br>heel | Patient's left<br>heel | Patient's right greater trochanter | Patient's left<br>greater<br>trochanter |
|---|---|---|---|---|---|
| SS1[N1] 2<br>SS1T[C34] | ○ Yes, likely to remain<br>assessable<br>○ Yes, unlikely to<br>remain assessable<br>○ No | Description (Control | | | 78 8 8 9 1 1 1 |
| Existing<br>pressure ulcer<br>on Day 1? | C Yes C No Category: | 0<br>0<br>0 0 0 0 | RE | FER TO SCREET | N 1.9 |
| s the body site<br>dry? | C Yes C No Type of moisture: ☐ Sweat ☐ Urine ☐ Diarrhea ☐ Other | | | List: 1<br>Variat | ion in audit trail:<br>to 5<br>ble: VARNAME<br>ion in export: |
| s the body site ntact? | C Yes C No | | | | ble: VARNAMEX |
| Are there dermatological contra-<br>ndications to apply dressing? | C Yes C No Skin condition: ☐ Incontinence- associated dermatitis ☐ Skin infection ☐ Other | | | | |
| s there any 1<br>ther contra-<br>ndication to<br>apply<br>dressing? | CYes CNo 2<br>OTHCI1[N1]<br>OTHCI1T[C3] | | | | |

| C Active support surface (such a | as alternating or low-air loss) |
|---|---|
| pressure redistributing) | in pressure dicers (standard roam, not |
| C Yes C No | |
| C At least every 2 hours | |
| C Every 3 - 4 hours | REFER TO SCREEN 1.9 |
| © Every 5 - 6 hours | |
| © Every 7 hours or more | |
| stionnaire | |
| 5L Quality of Life Questionnaire beer | n completed? C Yes C No |
| Patient | |
| Relative<br>Ward staff | |
| Other | |
| | ▼ |
| nne | |
| courantes | ▼ |
| | ▼ |
| ression | ▼ |
| té: (0 - 100) | |
| | Save Save and Next |
| | C Yes C No C At least every 2 hours C Every 3 - 4 hours C Every 5 - 6 hours C Every 7 hours or more stionnaire C Quality of Life Questionnaire been C Patient Relative Ward staff Other The Courantes |

#### 1.6.2. Droplists

#### Mobiliteit / Mobilité

# Dagelijkse activiteiten / Activités courantes

REFER TO SCREEN 1.9

Pijn, ongemak / Douleurs, gêne

Angst, somberheid / Anxiété, dépression

#### Zelfzorg / Autonomie de la personne

#### Category

I - Nonblanchable Erythema
II - Partial Thickness Skin Loss
III - Full Thickness Skin Loss
IV - Full Thickness Tissue Loss
Unstageable: Depth unknown
Suspected Deep Tissue Injury: Dept Unknown

# 1.7.1. Screen

| All answers must be checked "Yes" in order to be eligible for study participation | Von | No |
|---|---|---|
| | Yes | |
| <ol> <li>At risk for pressure ulcer development based on Braden risk assessment<br/>(Braden score ≤17).</li> </ol> | C | င |
| <ol> <li>Admitted to hospital within the previous 48 hours.</li> <li>Note: Not more than 25% of patients per site should be recruited at ICU wards.</li> </ol> | 0 | С |
| 3. Skin at sacrum is assessable and there is no clinically relevant incontinence-<br>associated dermatitis (IAD*) or another skin condition that would be a contra-<br>indication for the application of the devices under study, and there is no<br>pressure ulcer category II or worse present. | O | 0 |
| *clinically relevant IAD is defined as any of the 4 categories described in the publication<br>http://users.ugent.be/~dibeeckm/globiadnl/nlv1.0.pdf | | |
| 4. For at least 3 of the following 4 body sites (heel left, heel right, greater trochanter left greater trochanter right) one of the following two conditions should apply: | t, o | О. |
| <ul> <li>A study dressing can be applied as prevention of a pressure ulcer category II or worse at that body site (there is no contra-indication) OR</li> </ul> | | |
| - There is already a pressure ulcer category II or worse at that body site. | | |
| 5. Written informed consent by the patient or his/her legal representative. | О | 0 |
| Exclusion criteria | | |
| All answers must be checked "No" in order to be eligible for study participation | Yes | No |
| 1. Aged < 18 years. | 0 | 0 |
| <ol><li>The length of stay counting from first day of admission in one or (if the patient is<br/>transferred to another ward) more participating wards is &lt; 7 days.</li></ol> | С | О |
| 3. Both heels amputated | 0 | 0 |
| 4. Previously known/documented allergy for substances used in the devices under s | study. C | 0 |
| 5. A clinical condition not allowing participation in a clinical study. | 0 | C |
| 6. Participation in another interventional clinical trial. | 0 | 0 |
| <ol> <li>Patients who exceptionally receive or are planned to receive a dressing for the prevention of pressure ulcers at sacrum, heels and trochanters based on best medical judgment and outside of the surgery setting.</li> </ol> | С | c |
| Randomisation | | |
| Patient is randomised in arm: ARM[C16] | | |

Date of randomisation DENTRD[N2] DENTRM[N2] DENTRY[N4]

Time of randomisation TENTRH[N2] TENTRM[N2]

# 1.8. Day 1 - Study Intervention

# 1.8.1. Screen

PANEL = ASS

| | (dd) (mm) (yyyy) | Time: (hh on 24 hour clock) | |
|---|---|---|---|
| Is this day the end of slud | dy for this patient? | CYes CNo REFER T | O SCREEN 1.9 |
| 1. Ward Information | | | |
| Did the patient change w | ard since enrollment? | CYes CNo | |
| | | New ward type: OICU @ Non-IC | cu |
| 2. Study intervention | | 1 2 | ANYDRES[N1] |
| Has any silicone adhesiv | ve multilayer foam dressing b | | ANYDREST[C3] |
| | Dressing applied? | | |
| | Dressing applied? | Dressing type: | |
| Sacrum | CV CH | | |
| | C Yes C No | C Allever Life | |
| | DRESS1[N1] | ○ Allevyn® Life Sacrum<br>○ Allevyn® Life Heel | |
| | DRESS1T[C3] | C Mepilex® Border C Mepilex® Border Sacrum C Mepilex® Border Heel | 1= Ticked |
| | 1 | <ul> <li>Other silicone adhesive multila<br/>foam dressing</li> </ul> | ayer |
| | | Specify: | |
| Patient's right heel | C Yes C No | | |
| | O TES C NO | Ardinary none | |
| | | a feel flower arter and | |
| | DEEED TO | SCREEN 40 | |
| | REFER TO | SCREEN 1.9 | |
| Patient's left heel | REFER TO | SCREEN 1.9 | |
| Patient's left heel | REFER TO | THE THE PARTY | |
| Patient's left heel | | THE THE PARTY | Identification in audit trail: |
| Patient's left heel | | THE THE PARTY | List: 1 to 5 |
| Patient's left heel | | THE THE PARTY | List: 1 to 5<br>Variable: VARNAME |
| | | THE THE PARTY | List: 1 to 5 |
| Patient's right greater | | | List: 1 to 5<br>Variable: VARNAME<br>IPT: Dressing type |
| Patient's right greater | € Yes € No | | List: 1 to 5<br>Variable: VARNAME |
| Patient's right greater | € Yes € No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater | € Yes € No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater | € Yes € No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter | € Yes € No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's left heel Patient's right greater trochanter Patient's left greater trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter<br>Patient's left greater<br>trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |
| Patient's right greater<br>trochanter<br>Patient's left greater<br>trochanter | C Yes C No | | List: 1 to 5 Variable: VARNAME IPT: Dressing type Identification in export: |

# 1.9. Daily Assessment

# 1.9.1. Screen

PANEL = ASS

| | Daily Assessment | |
|---|---|---|
| DAY[C3]<br>1= Ticked | DAY Dale DDAYD[N2] DDAYD[N2] DDAYD[N1] DAYNA[N1] | |
| | Top I have been a | 1 2 te the last assessment? 1 CYes 2CNo WARDCH[N1] WARDCHT[C3] New ward type 1 CICU CNOHOU 2 WARDNEWIN1] WARDNEWTIC7] |
| | Adverse Device Effect / Devi Did any new Adverse Device Effe observed since last visit? | ect occour or was any new Device Deficiency Yes CNo 1 2 ADEDD[N1] ADEDDT[C3] |
| BR<br>BSEND[N1] | 4. Body sites evaluation | BRA3[N1] BRA4[N1] BRA5[N1] BRA6[N1] |
| 1= Ticked | Sacrum 1 Not Assessab | Heel right 2 Heel left 3 Greater 4 trochanter 5 Ite If Ticked: ASSESS1[N1] = 3 Identification in audit trail: ULCER1[N1] ULCER1T[C3] List: 1 to 5 |
| I=Sacrum<br>2=Heel right<br>3=Heel left | Photograph Cyes C No. | CAT1[N1] CAT1T[C42] Variable: VARNAME |
| = Greater trochanter riç<br>i=Greater trochanter le | ht 1 2 | PHOT1[N1] PHOT1T[C3] Identification in export: Variable: VARNAMEx |
| | hotograph taken of the pressure ucer category >= II developed during the study? | PHOULD1[N1] PHOULC1T[C3] |
| | is the body sit 2 1 Yes 2 No<br>dry? Type of moisture<br>Sweat | SWEAT1[N1] DARR1[N1] 1= Ticked |
| | Is the body site O'Yes O'No intact? | INTACT1[N1] INTACT1T[C3] |
| | Are there dematological Skin condition. contra- indications to apply dressing? G Yes S No of Skin condition. Skin infection. Skin infection. | INCONT [N1] |
| | Support information Support surface in bed. | 1 |
| | Heal(s) elevated from the bed?<br>Frequency of repositioning: | 1c Yes 2c No HEELELE[N1] HEELELET[C3] 1 c At least every 2 hours 2 c Every 3 - 4 hours 3 c Every 5 - 6 hours FREQREP[N1] FREQREPT[C22] 4 c Every 7 hours or more |

| | Has there been a c | hange of silicone | adhesive mu | ltilayer foam d | ressing since previous ass | essment? C Yes<br>1 | ®No CHDRES[N1]<br>2 | CHDREST C3 |
|---|---|---|---|---|---|---|---|---|
| | | Has there been<br>removal or<br>replacement or<br>placement at<br>this body site? | | y dressing<br>ed and not | Reason why dressing was replaced: | Reason why<br>dressing was newly<br>applied: | Dressing type applied<br>(enter the number applied<br>of each type): | |
| EN | Sacrum 1<br>2<br>REP1[N1]<br>REP1T[C12] | C No C Yes: Previous dressing removed 1 Replaced 2 Not replaced applied to the previously untreated body site | □ Body site assessa | egory >= 2 ogical n e no longer ble (bandage other medical | □ Saturated □ No longer fully adheres □ Dislodged □ Rolled at the edges □ Wrinkled □ Creased/damaged □ Soiled □ As per manufacturer's instructions □ Other | □ No contra-indications anymore □ Body site became treatable □ Other NAPNCI1[N1] NAPTREA1[N1] NAPOTH1[N1] 1= Ticked | □ Allevyn® Life □ Allevyn® Life Sacrum □ Allevyn® Life Heel □ Mepilex® Border □ Mepilex® Border Sacrum □ Mepilex® Border Heel □ Other silicone adhesive multilayer foam dressing Specify: | AL1[N1] ALS1[N1] ALH1[N1] MB1[N1] MBS1[N1] MBH1[N1] DRESOTH1[N |
| | CHANGE1<br>CHANGE1 | N1] | REMEC<br>REMUL<br>REMDE | | REPSAT1[N1]<br>REPNLA1[N1]<br>REPDISL1[N1] | | DRESOTS1[C255] | |
| 2 | Heel right | | REMNL<br>REMOT | | REPROLL1[N1]<br>REPWRIN1[N1] | | Identification in | audit trail: |
| 3 | Heel left | | 1= T | cked | REPSOIL1[N1] REPMAN1[N1] | | List: 1 to 5<br>Variable: V | ARNAME |
| | Greater<br>trochanter right | | | | REPOTH1[N1]<br>1= Ticked | | Identification in<br>Variable: V | |
| | Greater<br>trochanter left | | | | , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | | |
| | Н | conscious ST/<br>nconscious ST/<br>as the EQ - 5D - 5<br>ompleted by: 1 co | ATUS[N1 | ] STATU | • | | ] QOLCOMPT[C3] | |
| | Mobiliteit / Mobil | | | | | | OBIL[N1] MOBILT[ | |
| | and the second | mie de la personr<br>teiten / Activités c | | | | | UTONOM[N1] AUTO | |
| | Pijn, ongemak / I | | ourantes | | | | CTIVIT[N1] ACTIVI<br>AIN[N1] PAINT[C25 | |
| | | eid / Anxiété, dépre | ession | | | | EPRES[N1] DEPRI | |
| | Gezondheidsheid | dstoestand / Santé | é: [ | (0 - 1 | 00) HEALTH[A3] | | | |

#### 1.9.2. Droplists

#### Category \*

- 1 I Nonblanchable Erythema2 II Partial Thickness Skin Loss
- 3 III Full Thickness Skin Loss4 IV Full Thickness Tissue Loss

- 5 Unstageable: Depth unknown6 Suspected Deep Tissue Injury: Dept Unknown
- 8 II or higher classification unknown

#### Mobiliteit / Mobilité

Dagelijkse activiteiten / Activités courantes

Pijn, ongemak / Douleurs, gêne

Angst, somberheid / Anxiété, dépression

Zelfzorg / Autonomie de la personne

# 1.10. Termination

# 1.10.1. Screen

| | Termination |
|---|---|
| | Discontinuation of Study Intervention on ALL body sites |
| = TICKED | Date of end of study intervention on ALL body sites: (dd) (mm) (vvvv) |
| ENDDISC1[N1] | ☐ Non-compliance with study procedures |
| ENDDISC2[N1] | ☐ Life-threatening AE or Serious Adverse Event (SAE) that places the patient at immediate risk if the study intervention would be continued |
| ENDDISC3[N1] | Patient shows a worsening of his/her medical condition, which in the investigator's opinion requires a discontinuation of the study intervention |
| ENDDISC4[N1] | Patient's best interest |
| ENDDISC5[N1] | Contra-indications / inability to apply dressing on ALL body sites |
| ENDDISC6[N1] | Other Specify: ENDEXP6[C255] |
| | End of Study |
| | End of study date: (dd) (mm) (yyyy) DEOSD[N2] DEOSM[N2] DEOSY[N4] |
| = TICKED | Please indicate the reason for End of Study (check all that apply): |
| EOSDISC1[N1] | Patient is no longer at risk of pressure ulcer development according to the Braden scale (Braden score >17) |
| EOSDISC2[N1] | Day 14 reached |
| EOSDISC3[N1] | Patient withdrawal 1 2 |
| | Can collected data be kept in the study and used for the analysis? C Yes C No |
| EOSDISC4[N1] | Discharged from the hospital USEDATA[N1] USEDATAT[C3] |
| EOSDISC5[N1] | Moved to a non-participating ward |
| EOSDISC6[N1] | Death Date of death: (dd) (mm) (yyyy) |
| EOSDISC7[N1] | Study closure by sponsor DDTHD[N2] DDTHM[N2] DDTHY[N4] |
| EOSDISC8[N1] | Other |
| | Specify: EOSEXP8[C255] |
| | Back Save Save and Next |

# 1.11. Adverse Device Effects (ADE) Log

# 1.11.1. Screen

| Ξ | verse Device | Zirotto (i | | | | | | | A | dd |
|---|---|---|---|---|---|---|---|---|---|---|
| Nr | ADE descri | ption | Start Date<br>(dd/mm/yyyy) | Outcome | | esolved<br>n/yyyy) | Serious<br>ADE | Alerts | Monitor | a |
| | | | | | | | | | ja ja | X |
| AD | E number: | | ADENR[N | 13] | | | | | | |
| AD | E description: | Γ | ADENAME | E[C100] | | | | | | ia . |
| Se | verity: | 2 c<br>3 c | Mild AI<br>Moderate<br>Severe<br>NA/UK | DESEV[N1] | ADESEV | /T[C8] | | | | |
| Sta | art Date:<br>DADE | <br> SD[N2] | DADESM[N2] | DADESY[I | N4] | | | | | |
| Ou | tcome: | 1.0 | Resolved | | Date reso | olved: | | П | | |
| ΑĽ | DEOUT[N1] | ADEOUT | T[C8] | | DAI | DEED[A2 | DADEE | M[N2] | DADE | EY[N4] |
| | | 2 0 | Fatal | | Date of d | | (dd) | (mm) | (уууу) | |
| | | 3 6 | Ongoing | | DADED | THD[N2] | DADED | 1]MHT | N2] DAD | EDTHY |
| | | 4 0 | Unknown | | Date of la | ist assess | ment: (dd) | (mm) | (уууу) | |
| | rious ADE: | | Yes 2 o | ADESER | R[N1] AD | ESERT[ | | | l2] DAD | ELASY |
| Εv | ent considered | as: 10 | Expected 20 | | | | | 0] | | |
| | tion taken: | | | No ADEAC | | | | | | |
| = 7 | | | 1] □ Discontinu | | | | | cted bo | dy site(s) | 547 |
| | | | 1] Discontinu | | | n on ALL I | oody sites | | | |
| | ADE | EACT3[N | 1] □ Medication | n/Therapy | Specify: | ADEAG | CT3S[C25 | 5] | ^ | |
| | ADE | ACT4[N | 1] Other | | Specify: | | CT4S[C25 | | _ | |

# 1.12. Comments Log

# 1.12.1. Screen

| | Add comment | | | |
|---------|-------------|-----------------------|---------|---------|
| Nr | Screen | Comment | Alerts | Monitor |
| 100 | (m-50) | Otherwood performance | | × |
| Comme | ent number: | COMNR[N3] | | |
| Screen: | | COMSCR[C255] | | |
| Comme | ent | COMDES[C255] | rebar a | |
| | | , | | |
| | | 8 | | |
| | | y se " to se | | |
#### 1.13 Photographs Log

#### 1.13.1. Screen



### 1.14. Device Deficiency (DD) Log

#### 1.14.1. Screen

| _ | | | | | | | | Add |
|---|---|---|---|---|---|---|---|---|
| ۸r | DD description | Start Date<br>(dd/mm/yyyy) | End Date<br>(dd/mm/yyyy) | Related to (S)ADE | Alerts | Monitor | | |
| | | | 10 | | | | X | |
| | Date: | | DDDSY[N4] | licable / Unkr | nown [ | DDNA[N1 | i] DD | NAT[C24] |
| | DDDED[A2 | (dd) (mm) (yyyy<br>2] DDDEM[N2] | 1 O Not App<br>)<br>DDDEY[N4] | | nown [ | DDNA[N1 | ] DD | NAT[C24] |
| Rek | ated to an (S)ADE: 1<br>DDREL[N1 | OYes 201<br>] DDRELT[C3] | | number(s): | | | DDAD | ENR[C35] |

#### 1.15. Investigator Statement

#### 1.15.1. Screen

| | Investigator Sta | atement | | | | | PA | NEL = ( | GEN |
|---|---|---|---|---|---|---|---|---|---|
| | INV[N1] | | | | 7 | | | | |
| = TICKED | ☐ By signing I ce<br>have been rev | ertify that the data in<br>iewed by a medic | reported in the eal doctor. | eCRF are accura | te and comp | olete and t | that all saf | ety related | d data |
| | | | | | | | | | 1.1 |
| | User ID: | | | | | | | | 8 |
| | | | | | | | | | 0.0 |
| | Password: | | | (4) | | | | | |
| | Back | | | | | | | Sa | wa 1 |





### APPENDIX 2. TEMPLATE TABLES RESULTS (1) PATIENT INFO

Table 1. Patient's baseline demographics (categorical variables), by Randomised Arm, ITT population

| | | | Rando | mised arm | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | llevyn<br>Life® | | epilex<br>rder® | | dard of<br>Care | | Γotal |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Consent signed by | | | | | | | | |
| Patient | 1 | 25.0 % | 2 | 40.0 % | 1 | 100.0 % | 4 | 40.0 % |
| Legal representative | 3 | 75.0 % | | | 0 | 0 | 6 | 60.0 % |
| Ward type on which patient is staying (corrected) | | | | | | | | |
| ICU | 0 | | 1 | 20.0 % | Ь | 0 | 1 | 10.0 % |
| Non-ICU | 4 | % | 4 | 80.0 | 1 | 100.0 % | 9 | 90.0 % |
| Age (years) | | | | | | | | |
| <60 | 0 | 0 | | J.0 % | 0 | 0 | 1 | 10.0 % |
| 60-69 | 0 | 0 | | 2,0 % | 0 | 0 | 1 | 10.0 % |
| 70-79 | 3 | 0 | 2 | | 0 | 0 | 2 | 20.0 % |
| >=80 | 7. | 0/2 | 1 | 20.6 | 1 | 100.0 % | 6 | 60.0 % |
| Gender type | | | | | | | | |
| Female | 4 | .0 % | 4 | J.0 % | 1 | 100.0 % | 9 | 90.0 % |
| Male | | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| wii_cat | | | | | | | | |
| Normal weigh | | 100.0 % | 2 | 40.0 % | 1 | 100.0 % | 7 | 70.0 % |
| Overweight | | 0 | 2 | 40.0 % | 0 | 0 | 2 | 20.0 % |
| Obesity | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| type | | | | | | | | |
| No | 4 | 100.0 % | 2 | 40.0 % | 1 | 100.0 % | 7 | 70.0 % |
| Yes | 0 | 0 | 3 | 60.0 % | 0 | 0 | 3 | 30.0 % |
| Expected sta, | | | | | | | | |
| 7 days or more | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Surgery type | | | | | | | | |
| No | 3 | 75.0 % | 5 | 100.0 % | 1 | 100.0 % | 9 | 90.0 % |
| Yes | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| Type of surgery | | | | | | | | |
| 3. 3. | 3 | 75.0 % | 5 | 100.0 % | 1 | 100.0 % | 9 | 90.0 % |
| Non-elective | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| Anaesthesia type | | | | | | | | |
| | 3 | 75.0 % | 5 | 100.0 % | 1 | 100.0 % | 9 | 90.0 % |
| General | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |

Table 2. Inclusion and Exclusion Criteria, by Randomised Arm, ITT population

| | | | Rando | mised arm | | | | |
|---|---|---|---|---|---|---|---|---|
| | | levyn<br>.ife® | | epilex<br>rder® | | dard of<br>are | - | Γotal |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Inclusion criteria 1 | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Inclusion criteria 2 | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Inclusion criteria 3 | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100.0 % | | | 10 | 100.0 % |
| Inclusion criteria 4 | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 10 | 1 | 100.0 % | | 100.0 % |
| Inclusion criteria 5 | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100. | 1 | 10 | 10 | 100.0 % |
| Exclusion criteria 1 | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | | 90.0 % | 10 | 100.0 % |
| Exclusion criteria 2 | • | | | | | | | |
| No | 4 | 2 % | | 0 % | 1 | 100. | 10 | 100.0 % |
| Exclusion criteria 3 | | | | | | | | |
| No | 4 | 100. | 5 | % | | 3 % | 10 | 100.0 % |
| Exclusion criteria 4 | | | | | | | | |
| No | 4 | 100.0 % | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| sion criteria 5 | | Ì | | | | | | |
| | | 20% | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| clusion cris | | | 1 | | | | | |
| | 4 | 100 | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Exclusion criteria 7 | | | | | | | | |
| No | 4 | % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |

Table 3. Patient's baseline demographics (continuous variables), by Randomised Arm, ITT population

| | | R | andomised a | arm | |
|---|---|---|---|---|---|
| | | Allevyn<br>Life® | Mepilex<br>Border® | Standard of Care | Total |
| Age (years) | N | 4 | 5 | 1 | 10 |
| | Mean | 84.2 | 73.1 | 91.2 | 79.3 |
| | Std | 3.2 | 9.4 | 0 | 9.5 |
| | Min | 80.5 | 59.2 | 91.2 | 59.2 |
| | Q1 | 82.0 | 69.6 | 91.2 | 74.3 |
| | Median | 84.2 | 74.3 | 91.2 | 82.0 |
| | Q3 | | 78.1 | 91.2 | 84.8 |
| | | 86 | 84.0 | 91.2 | 91.2 |
| | Miss | 0 | 0 | 0 | 0 |
| Braden score (code) | N | 4 | 5 | 1 | 10 |
| | ean | | 12.6 | 17.0 | 12.4 |
| | | 0.8 | 2.3 | 0 | 2.4 |
| | Min | 10.0 | 11.0 | 17.0 | 10.0 |
| | Q1 | 5 | 11.0 | 17.0 | 11.0 |
| | Median | | 11.0 | 17.0 | 11.0 |
| | | 11.5 | 14.0 | 17.0 | 14.0 |
| | Max | 12.0 | 16.0 | 17.0 | 17.0 |
| | NMiss | 0 | 0 | 0 | 0 |
| Time (days) between angery and informed conse | N | 1 | 0 | 0 | 1 |
| | Mean | 2.0 | 0 | 0 | 2.0 |
| | Std | 0 | 0 | 0 | 0 |
| | Min | 2.0 | 0 | 0 | 2.0 |
| | Q1 | 2.0 | 0 | 0 | 2.0 |
| | Median | 2.0 | 0 | 0 | 2.0 |
| | Q3 | 2.0 | 0 | 0 | 2.0 |
| | Max | 2.0 | 0 | 0 | 2.0 |
| | NMiss | 3 | 5 | 1 | 9 |

Table 3. Patient's baseline demographics (continuous variables), by Randomised Arm, ITT population

| | | R | andomised | arm | |
|---|---|---|---|---|---|
| | | Allevyn<br>Life® | Mepilex<br>Border® | Standard of Care | Total |
| Time (days) between hosp admission and informed consent | N | 4 | 5 | 1 | 10 |
| | Mean | 2.0 | 1.8 | 2.0 | 1.9 |
| | Std | 0.8 | 0.4 | 0 | 0.6 |
| | Min | 1.0 | 1.0 | 2.0 | 1.0 |
| | Q1 | 1.5 | 2.0 | 2.0 | 2.0 |
| | Median | 2.0 | 2.0 | 2.0 | 2.0 |
| | Q3 | | 2.0 | 2.0 | 2.0 |
| | | 3. | 2.0 | 2.0 | 3.0 |
| | Miss | 0 | 0 | 0 | 0 |
| Time (days) between informed consent and randomisat | N | A | 5 | 1 | 10 |
| | ean | | 1.0 | 1.0 | 1.0 |
| | | 0.0 | 0.0 | 0 | 0.0 |
| | Min | 1.0 | 1.0 | 1.0 | 1.0 |
| | Q1 | | 1.0 | 1.0 | 1.0 |
| | Median | | 1.0 | 1.0 | 1.0 |
| | | 1.0 | 1.0 | 1.0 | 1.0 |
| | Max | 1.0 | 1.0 | 1.0 | 1.0 |
| | NMiss | 0 | 0 | 0 | 0 |
| Time (days) between andomisation and termination | N | 4 | 5 | 0 | 9 |
| | Mean | 13.3 | 9.2 | 0 | 11.0 |
| | Std | 1.5 | 3.1 | 0 | 3.2 |
| | Min | 12.0 | 6.0 | 0 | 6.0 |
| | Q1 | 12.0 | 7.0 | 0 | 9.0 |
| | Median | 13.0 | 9.0 | 0 | 12.0 |
| | Q3 | 14.5 | 10.0 | 0 | 14.0 |
| | Max | 15.0 | 14.0 | 0 | 15.0 |
| | NMiss | 0 | 0 | 1 | 1 |

Table 3. Patient's baseline demographics (continuous variables), by Randomised Arm, ITT population

| | | R | andomised a | arm | |
|---|---|---|---|---|---|
| | | Allevyn<br>Life® | Mepilex<br>Border® | Standard of Care | Total |
| Time (days) between randomisation and end of study | N | 4 | 5 | 1 | 10 |
| | Mean | 13.3 | 9.2 | 8.0 | 10.7 |
| | Std | 1.5 | 3.1 | 0 | 3.2 |
| | Min | 12.0 | 6.0 | 8.0 | 6.0 |
| | Q1 | 12.0 | 7.0 | 8.0 | 8.0 |
| | Median | 13.0 | 9.0 | 8.0 | 11.0 |
| | Q3 | | 10.0 | 8.0 | 14.0 |
| | | 16 | 14.0 | 8.0 | 15.0 |
| | Miss | 0 | 0 | 0 | 0 |
| Body Mass Index | N | 4 | 5 | 1 | 10 |
| | ean | | 28.7 | 24.6 | 25.5 |
| | | 1.4 | 9.8 | 0 | 7.5 |
| | Min | 20.3 | 23.4 | 24.6 | 20.3 |
| | Q1 | ę | 23.4 | 24.6 | 22.0 |
| | Median | 2 | 25.0 | 24.6 | 23.4 |
| | | 22.7 | 25.6 | 24.6 | 25.0 |
| | Max | 23.4 | 46.1 | 24.6 | 46.1 |
| | NMiss | 0 | 0 | 0 | 0 |
| Height (cm) | N | 4 | 5 | 1 | 10 |
| | Mean | 159.3 | 158.2 | 165.0 | 159.3 |
| | Std | 8.6 | 2.0 | 0 | 5.6 |
| | Min | 149.0 | 155.0 | 165.0 | 149.0 |
| | Q1 | 153.5 | 158.0 | 165.0 | 158.0 |
| | Median | 159.0 | 158.0 | 165.0 | 159.0 |
| | Q3 | 165.0 | 160.0 | 165.0 | 160.0 |
| | Max | 170.0 | 160.0 | 165.0 | 170.0 |
| | NMiss | 0 | 0 | 0 | 0 |

Table 3. Patient's baseline demographics (continuous variables), by Randomised Arm, ITT population

| | | R | andomised | arm | |
|---|---|---|---|---|---|
| | | Allevyn<br>Life® | Mepilex<br>Border® | Standard of Care | Total |
| Weight (kg) | N | 4 | 5 | 1 | 10 |
| | Mean | 54.8 | 71.8 | 67.0 | 64.5 |
| | Std | 3.8 | 24.2 | 0 | 18.4 |
| | Min | 52.0 | 60.0 | 67.0 | 52.0 |
| | Q1 | 52.0 | 60.0 | 67.0 | 55.0 |
| | Median | 53.5 | 60.0 | 67.0 | 60.0 |
| | Q3 | | 64.0 | 67.0 | 64.0 |
| | | 64 | 115.0 | 67.0 | 115.0 |
| | Miss | 0 | 0 | 0 | 0 |



Table 4. Braden scale at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arn | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | levyn<br>.ife® | | epilex<br>rder® | | dard of<br>are | - | Γotal |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| BRADEN_cat | | | | | | | | |
| 10-14 | 4 | 100.0 % | 4 | 80.0 % | 0 | 0 | 8 | 80.0 % |
| 15-19 | 0 | 0 | 1 | 20.0 % | 1 | 100.0 % | 2 | 20.0 % |
| Braden scale assessement - Sensory (code) | | | | | | | | |
| 2 | 2 | 50.0 % | 2 | 40.0.% | 0 | 0 | 4 | 40.0 % |
| 3 | 2 | 50.0 % | 1 | | | 0 | 3 | 30.0 % |
| 4 | 0 | 0 | | 40.0 % | | 100.0 % | 3 | 30.0 % |
| Braden scale assessement - Moisture (code) | | | | | | | | |
| 1 | 0 | | 1 | 20.0 % | | 0 | 1 | 10.0 % |
| 2 | 3 | 75.0 % | | 40.0 % | 1 | 0 | 5 | 50.0 % |
| 3 | 1 | 25.0 % | 2 | | 1 | 100.0 % | 4 | 40.0 % |
| Braden scale assessement - Activity (code) | | | | | | | | |
| 1 | | 75.0 % | 2 | 40. | 0 | 0 | 5 | 50.0 % |
| 2 | 1 | | 3 | 60.0 % | | 100.0 % | 5 | 50.0 % |
| Braden scale assessement - Mobility (cod | | | | | | | | |
| 1 | | 25.6 | 0 | | 0 | 0 | 1 | 10.0 % |
| 2 | | % | 4 | 80.0 % | 0 | 0 | 7 | 70.0 % |
| 3 | | 0 | 1 | 20.0 % | 1 | 100.0 % | 2 | 20.0 % |
| Braden scale essement - Nutrition (code) | | | | | | | | |
| 1 | 1 | ρ % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| 2 | 3 | % | 4 | 80.0 % | 0 | 0 | 7 | 70.0 % |
| 3 | О | 0 | 1 | 20.0 % | 1 | 100.0 % | 2 | 20.0 % |
| Braden scale assessement - Friction (code | | | | | | | | |
| 1 | 2 | 50.0 % | 3 | 60.0 % | 0 | 0 | 5 | 50.0 % |
| 2 | 2 | 50.0 % | 2 | 40.0 % | 1 | 100.0 % | 5 | 50.0 % |



Table 5a. Sacrum evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arn | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | llevyn<br>_ife® | | epilex<br>rder® | | dard of<br>Care | | Total |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Body site assessable type - Sacrum | | | | | | | | |
| Yes, likely to remain assessable | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Presence of pressure ulcer - Sacrum | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Category - Sacrum (code) | | | | | | | | |
| | 4 | 100.0 % | | | 1 | 100.0 % | 10 | 100.0 % |
| Photograph taken - Sacrum | | | | | | | | |
| | 4 | /6 | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Photo taken category >= II - Sacrum | | | | | | | | |
| | 4 | 16 | 5 | 1 10 | 1 | 100.0 % | 10 | 100.0 % |
| Is the body site dry - Sacrum | | | | | | | | |
| No | 1 | 25.0 % | | 20.0 % | 0 | 0 | 2 | 20.0 % |
| Yes | 3 | 75.0 % | 4 | % | 1 | 100.0 % | 8 | 80.0 % |
| Type of moisture - Sweat - Sacrum (cod | | | | | | | | |
| | 4 | | 5 | 100.0 5 | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Urine - Sacrum (code) | | | | | | | | |
| | | 75.0 % | 5 | 100.0 % | 1 | 100.0 % | 9 | 90.0 % |
| 1 | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| Type of moir - Diarrhea - Sacrum (code) | | | | | | | | |
| | | 100.0 % | 4 | 80.0 % | 1 | 100.0 % | 9 | 90.0 % |
| 1 | | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Type of mo Sacrum (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is body site intact - Sacrum | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Dermatologic contra-indications - Sacrum | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - incontience-associated - Sacrum (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Skin infection - Sacrum (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Other - Sacrum | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |



Table 5a. Sacrum evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arm | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | Allevyn<br>Life® | | | | Standard of<br>Care | | - | Total |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Is there other contra-indication - Sacrum | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |



Table 5b. Heel right evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | omised arm | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | levyn<br>Life® | | epilex<br>order® | | idard of<br>Care | | Total |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Body site assessable type - Heel right | | | | | | | | |
| Yes, likely to remain assessable | 3 | 75.0 % | 5 | 100.0 % | 1 | 100.0 % | 9 | 90.0 % |
| Yes, unlikely to remain assessable | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| Presence of pressure ulcer - Heel right | | | | | | | | |
| | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| No | 3 | 75.0 % | | | 1 | 100.0 % | 8 | 80.0 % |
| Yes | 0 | | 1 | 20.0 | 0 | 0 | 1 | 10.0 % |
| Category - Heel right (code) | | | | | | | | |
| | 4 | 0 % | 4 | 80 | 1 | 100.0 % | 9 | 90.0 % |
| III - Full Thickness Skin Loss | 0 | | 1 | //0 | 0 | 0 | 1 | 10.0 % |
| Photograph taken - Heel right | | | | | | | | |
| | 4 | 100.0 % | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Photo taken category >= II - Heel rig | | | | | | | | |
| | | 100.0 % | 5 | | 1 | 100.0 % | 10 | 100.0 % |
| Is the body site dry - Heel right | | | | | | | | |
| | 1 | ٥.0 % | | 0 | 0 | 0 | 1 | 10.0 % |
| No | | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Yes | 3 | 75.0 % | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |
| Type of moi - Sweat - Heel right (code) | | | | | | | | |
| | | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of n ure - Urine and (Coc. | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Diarrhea - Heel right (cod | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Oth | | | | | | | | |
| | 4 | 100.0 % | 4 | 80.0 % | 1 | 100.0 % | 9 | 90.0 % |
| 1 | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Is body site intact - Heel right | | | | | | | | |
| | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| No | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Yes | 3 | 75.0 % | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |
| Dermatologic contra-indications - Heel right | | | | | | | | |
| | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| No | 3 | 75.0 % | 5 | 100.0 % | 1 | 100.0 % | 9 | 90.0 % |

Table 5b. Heel right evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arm | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | Allevyn<br>Life® | | epilex<br>rder® | | dard of<br>are | - | Total |
| | N | N Col % | | Col % | N | Col % | N | Col % |
| Skin condition - incontience-associated - Heel right (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Skin infection - Heel right (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Other - Heel right | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is there other contra-indication - Heel right | | | | | | | | |
| | 1 | 25.0 | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| No | 3 | /0 | 5 | 100.0 | 1 | 100.0 % | 9 | 90.0 % |



Table 5c. Heel left evaluation at Day 1, by Randomised Arm, ITT population

| | | llevyn<br>_ife® | | epilex<br>rder® | | dard of<br>Care | | Total |
|---|---|---|---|---|---|---|---|---|
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Body site assessable type - Heel left | | | | | | | | |
| Yes, likely to remain assessable | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Presence of pressure ulcer - Heel left | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Category - Heel left (code) | | | | | | | | |
| | 4 | 100.0 % | | | 1 | 100.0 % | 10 | 100.0 % |
| Photograph taken - Heel left | | | | | | | | |
| | 4 | //0 | 5 | 100.0 9 | 1 | 100.0 % | 10 | 100.0 % |
| Photo taken category >= II - Heel left | | | | | | | | |
| | 4 | 16 | 5 | //0 | 1 | 100.0 % | 10 | 100.0 % |
| Is the body site dry - Heel left | | | | | | | | |
| Yes | 4 | 100.0 % | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Sweat - Heel left (o | | | | | | | | |
| | | 20.0 % | 5 | 16 | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Urine - Heel left (code) | | | | | | | | |
| | 4 | J.0 % | | 0.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Diarrhea - Heel left (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of mg s - Other - Heel left (code) | | | | | | | | |
| | | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is v site intact | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Dermatologic contra-indications - Heel lef | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - incontience-a | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Skin infection - Heel left (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Other - Heel left | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is there other contra-indication - Heel left | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |

Table 5d. Greater trochanter right evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arn | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | llevyn<br>Life® | | epilex<br>rder® | | dard of<br>Care | | Total |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Body site assessable type - Greater trochanter right | | | | | | | | |
| Yes, likely to remain assessable | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Presence of pressure ulcer - Greater trochanter right | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Category - Greater trochanter right (code) | | | | | | | | |
| | 4 | | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Photograph taken - Greater trochanter right | | | | | | | | |
| | | 100.0 % | 5 | .0 % | 1 | 100.0 % | 10 | 100.0 % |
| Photo taken category >= II - Greater trochanter right | | | | | | | | |
| | | 100.0 % | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is the body site dry - Greater trochanter right | | | | | | | | |
| Yes | 4 | 16. | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Sweat - Greater trochanter | | | | | | | | |
| | 4 | 100.0 % | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Urine - Greater trochanter right | • | | | | | | | |
| | 4 | 10 | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Diarrhea - Greater trochanter right | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture Greater trochanter right (code | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is body sit tact - Great the right | | | | | | | | |
| Yes | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Dermatologic contra-indications - Greater trochan | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - incontience-associate and anter right (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Skin infection - Greater trochanter right (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Other - Greater trochanter right | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is there other contra-indication - Greater trochanter right | | | | | | | | |
| No | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |



Table 5e. Greater trochanter left evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arn | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | llevyn<br>Life® | | epilex<br>order® | | dard of<br>Care | - | Total |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Body site assessable type - Greater trochanter left | | | | | | | | |
| No | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| Yes, likely to remain assessable | 3 | 75.0 % | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |
| Yes, unlikely to remain assessable | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Presence of pressure ulcer - Greater trochanter left | | | | | | | | |
| | 1 | 2 | | 20.0 % | 0 | 0 | 2 | 20.0 % |
| No | 3 | .0 % | 4 | 0 % | 1 | 100.0 % | 8 | 80.0 % |
| Category - Greater trochanter left (code) | | | | | | | | |
| | | 100.0 % | 5 | 0.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Photograph taken - Greater trochanter left | | | 4 | | | | | |
| | 4 | | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Photo taken category >= II - Greater trochanter left | | • | | | | | | |
| | 4 | 100.0 % | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is the body site dry - Greater trochanter | | | | | | | | |
| | | % | 1 | 20.0 % | 0 | 0 | 2 | 20.0 % |
| Yes | | 10. | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |
| Type of moisture - Sweat - Greater trochanter left (c | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture e - Greater trochanter left (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture rrhea - Groger anter pde) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Type of moisture - Other - Greater trochanter left | - | | | | - | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is body site intact - Gr | • | 10010 70 | | 100.0 /6 | | 10010 70 | | .00.0 /0 |
| io body one intakt on | 1 | 25.0 % | 1 | 20.0 % | 0 | 0 | 2 | 20.0 % |
| Yes | 3 | 75.0 % | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |
| Dermatologic contra-indications - Greater trochanter left | | 70.0 70 | т . | 00.0 70 | • | 100.0 70 | | 00.0 /0 |
| 25. matologio contra malocalorio - Gioder trochanter lett | 1 | 25.0 % | 1 | 20.0 % | 0 | 0 | 2 | 20.0 % |
| No | 3 | 75.0 % | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |
| Skin condition - incontience-associated - Greater trochanter left (code) | 3 | 7 3.0 70 | - | 00.0 /0 | ı | 100.0 /0 | U | 00.0 /0 |
| OKIN CONGRESION - INCOMMENCE-associated - Greater trochlanter left (code) | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Skin condition - Skin infaction - Greater trachenter left (and a) | 4 | 100.0 % | ວ | 100.0 % | - | 100.0 % | 10 | 100.0 % |
| Skin condition - Skin infection - Greater trochanter left (code) | | 100.0.0/ | _ | 100.0.00 | 4 | 100.0.07 | 40 | 100.00/ |
| • | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |

Table 5e. Greater trochanter left evaluation at Day 1, by Randomised Arm, ITT population

| | | | Rando | mised arm | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | Allevyn<br>Life® | | Mepilex<br>Border® | | | dard of<br>are | | Total |
| | N Col % | | N Col % | | N Col % | | N | Col % |
| Skin condition - Other - Greater trochanter left | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Is there other contra-indication - Greater trochanter left | | | | | | | | |
| | 1 | 25.0 % | 1 | 20.0 % | 0 | 0 | 2 | 20.0 % |
| No | 3 | 75.0 % | 4 | 80.0 % | 1 | 100.0 % | 8 | 80.0 % |



Table 6. Support information at Day 1, by Randomised Arm, ITT population

| | | Allevyn<br>Life® | | epilex<br>order® | | dard of<br>are | | |
|---|---|---|---|---|---|---|---|---|
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0<br>% | 5 | 100.0<br>% | 1 | 100.0<br>% | 10 | 100.0<br>% |
| Support information type | | | | | | 100.0 | | |
| Active support surface (such as alternating or low-air loss) | 0 | 0 | 1 | 20.0 % | 1 | % | 2 | 20.0 % |
| No specific mattress to prevent pressure ulcers (standard foam, not pressure redistributing) | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Reactive support surface (such as visco-elastic foam or air-filled) | 1 | 100.0 | 3 | 60.0 % | 0 | 0 | 7 | 70.0 % |
| Heels elevated from bed | | | | | | | | |
| No | 3 | 75.0 % | | 60.0 % | 0 | 0 | 6 | 60.0 % |
| Yes | 1 | 25.0 9 | 2 | 40.0 % | 1 | 100.0<br>% | 4 | 40.0 % |
| Frequency of repositioning type | | | | | | 100.0 | | |
| Every 3-4 hours | | .0 % | 1 | 20.0 % | 1 | % | 4 | 40.0 % |
| Every 5-6 hours | 2 | 0 % | 2 | 40.0 % | 0 | 0 | 4 | 40.0 % |
| Every 7 hours or more | 0 | | 2 | 40.0 % | 0 | 0 | 2 | 20.0 % |



Table 2. Pressure Ulcer and Randomised Arm, by anatomic site

| | | | Rando | mised arm | 1 | | | |
|---|---|---|---|---|---|---|---|---|
| | | levyn<br>.ife® | | epilex<br>order® | | dard of<br>Care | - | Γotal |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Total | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for discontinuation-Non compliance (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for discontinuation-Life threatening AE or SAE (code) | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for discontinuation-Worsening medical condition (code) | | | | | | | | |
| | 4 | 100.0 | | 2 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for discontinuation-Patient's best interest (code) | | | | | | | | |
| | 4 | 0.0 % | 5 | 10 | 1 | 100.0 % | 10 | 100.0 % |
| Reason for discontinuation-Contra indications (code) | | | | | | | | |
| | 4 | 2 % | 5 | 0.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Other reasons for discontinuation (code) | | | 47 | | | | | |
| | 0 | 0 | | 0 | 1 | 100.0 % | 1 | 10.0 % |
| 1 | 4 | 100.0 % | | 100.0 % | 0 | 0 | 9 | 90.0 % |
| Other reasons to discontinue | | | | | | | | |
| | 6 | | 0 | 0 | 1 | 100.0 % | 1 | 10.0 % |
| DAY 14 REACHED | | 0 | | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Discharged from the hospital | 2 | 50.0 % | 0 | 0 | 0 | 0 | 2 | 20.0 % |
| EOS (day 14 reached) | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| End of study (day 14 re 4) | 1 | 25.0 % | 0 | 0 | 0 | 0 | 1 | 10.0 % |
| death | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| discharged | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| no longer at risk | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| ontslag uit ziekenhuis | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Reason for end of study - no risk of pressy | | | | | | | | |
| | 4 | 100.0 % | 4 | 80.0 % | 0 | 0 | 8 | 80.0 % |
| 1 | 0 | 0 | 1 | 20.0 % | 1 | 100.0 % | 2 | 20.0 % |
| Reason for end of study - Day 14 reached | | | | | | | | |
| | 2 | 50.0 % | 4 | 80.0 % | 1 | 100.0 % | 7 | 70.0 % |
| 1 | 2 | 50.0 % | 1 | 20.0 % | 0 | 0 | 3 | 30.0 % |
| Reason for end of study - Patient withdraw | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for end of study - Discharged from hospital | | | _ | | | | | |
| | 2 | 50.0 % | 3 | 60.0 % | 1 | 100.0 % | 6 | 60.0 % |
| 1 | 2 | 50.0 % | 2 | 40.0 % | 0 | 0 | 4 | 40.0 % |

Table 2. Pressure Ulcer and Randomised Arm, by anatomic site

| | Randomised arm | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Allevyn<br>Life® | | Mepilex<br>Border® | | Standard of<br>Care | | | Total |
| | N | Col % | N | Col % | N | Col % | N | Col % |
| Reason for end of study - Moving to non-participating ward | | | | | | | | |
| | 4 | 100.0 % | 5 | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for end of study - Death | | | | | | | | |
| | 4 | 100.0 % | 4 | 80.0 % | 1 | 100.0 % | 9 | 90.0 % |
| 1 | 0 | 0 | 1 | 20.0 % | 0 | 0 | 1 | 10.0 % |
| Reason for end of study - Study closure by sponsor (code) | | | | | | | | |
| | 4 | 100.0 | | Q % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for end of study - Other (code) | | | | | | | | |
| | 4 | 0.0 % | 5 | 10 | 1 | 100.0 % | 10 | 100.0 % |
| Collected data can be used for the analysis type | | | | | | | | |
| | 4 | 0 % | 5 | J.0 % | 1 | 100.0 % | 10 | 100.0 % |
| Reason for end of study - Other | | | | | | | | |
| _ | 4 | 100.0 | | 100.0 % | 1 | 100.0 % | 10 | 100.0 % |



### **APPENDIX 3. TEMPLATE TABLES RESULTS (2) CLINICAL OUTCOMES**

Table 1. Patient's characteristics, by Pressure Ulcer

| | | Pressu | | | | |
|---|---|---|---|---|---|---|
| | , | Yes | | No | T | otal |
| | N | % | N | % | N | % |
| Total | 2 | 20.0 | 8 | 80.0 | 10 | 100.0 |
| Site | | | | | | |
| AZ Groeninge | | 0.0 | | 0.00 | 4 | 100.0 |
| UZ Brussel | U | 0.0 | 1 | 0.0 | 1 | 100.0 |
| Aalst | 1 | 50.0 | 1 | 0.0 | 2 | 100.0 |
| AZ Zottegem | 0 | 0.0 | | 100.0 | 1 | 100.0 |
| UZ Leuven | | 1 | 0 | 0.0 | 1 | 100.0 |
| OLV Waregem | 0 | | 1 | 100.0 | 1 | 100.0 |
| Age (yea | | | | | | |
| <60 | 0 | 0.0 | | 0.00 | 1 | 100.0 |
| 60-69 | | 20 | 1 | 100.0 | 1 | 100.0 |
| 70-79 | 0 | | 2 | 100.0 | 2 | 100.0 |
| >=80 | 2 | 33.3 | 4 | 66.7 | 6 | 100.0 |
| Gender type | | | | | | |
| Fema | 2 | 22.2 | 7 | 77.8 | 9 | 100.0 |
| Male | 0 | 0.0 | 1 | 100.0 | 1 | 100.0 |
| BMI_cat | | | | | | |
| Normal weight | 2 | 28.6 | 5 | 71.4 | 7 | 100.0 |
| Overweight | 0 | 0.0 | 2 | 100.0 | 2 | 100.0 |
| Obesity | 0 | 0.0 | 1 | 100.0 | 1 | 100.0 |
| Diabete type | | | | | - | |
| No | 2 | 28.6 | 5 | 71.4 | 7 | 100.0 |
| Yes | 0 | 0.0 | 3 | 100.0 | 3 | 100.0 |
| Ward type on which patient is staying (corrected) | | | | | | |
| ICU | 0 | 0.0 | 1 | 100.0 | 1 | 100.0 |
| Non-ICU | 2 | 22.2 | 7 | 77.8 | 9 | 100.0 |

Table 2. Pressure Ulcer and Randomised Arm, by anatomic site

| | | Pressu | re u | lcer | | |
|------------|---|--------|------|-------|---|-------|
| | | Yes | | No | T | otal |
| | N | N % | | % | N | % |
| BRADEN_cat | | | | | | |
| 10-14 | 2 | 25.0 | 6 | 75.0 | 8 | 100.0 |
| 15-19 | 0 | 0.0 | 2 | 100.0 | 2 | 100.0 |

| | | Randomi | ised ar | m | | |
|---|---|---|---|---|---|---|
| | Trea | atment | | dard of<br>are | | Γotal |
| | N | Col | N | Col | N | Col |
| Total | 9 | 100.00 | 1 | 100.00 | 10 | 100 |
| PU All sites | | | | | | |
| Yes | 2 | 22.22 | 0 | 0.00 | | 0.00 |
| No | 7 | 77.78 | 1 | 100.00 | 8 | |
| PU Sacrum | | | | | | |
| Yes | 2 | 22.22 | | 0.00 | 2 | 20.00 |
| No | 7 | 77.78 | | | 8 | 80.00 |
| PU Heel R | | | | | | |
| • | 1 | 11.11 | 0 | 0.00 | 1 | )<br>2 <b>A</b> |
| Yes | 0 | 0.00 | 0 | 00 | | 0.00 |
| No | | .89 | 1 | 1 | 9 | 90.00 |
| PU H | | | | | | |
| Yes | 0 | 0.0 | | 0.0 | 6 | 0.00 |
| No | 0 | .010 | | 00.00 | 10 | 100.00 |
| PU Tro | | | | | | |
| Yes | 0 | 0.00 | 9 | 0.00 | 0 | 0.00 |
| No | 9 | 100.00 | | 100.00 | 10 | 100.00 |
| PU Troch L | | | | | | |
| Yes | 0 | 0.00 | 0 | 0.00 | 0 | 0.00 |
| No | 9 | 100.00 | 1 | 100.00 | 10 | 100.00 |

Table 2. Pressure Ulcer and Randomised Arm, by anatomic site

| | | R | ando | mised ar | m | | | |
|---|---|---|---|---|---|---|---|---|
| | | levyn<br>.ife® | | pilex<br>rder® | | dard of<br>are | - | Γotal |
| | N | Col | N | Col | N | Col | N | Col |
| Total | 4 | 100.00 | 5 | 100.00 | 1 | 100.00 | 10 | 100.00 |
| PU All sites | | | | | | | | |
| Yes | 2 | 50.00 | 0 | 0.00 | 0 | 0.00 | 2 | 20.00 |
| No | 2 | 50.00 | 5 | 100.00 | 1 | 100.00 | 8 | 80.00 |
| PU Sacrum | | | | | | | | |
| Yes | 2 | 50.00 | 0 | 0.00 | 0 | | 0 | 20.00 |
| No | 2 | 50.00 | 5 | 100.00 | | 100.00 | | 80.00 |
| PU Heel R | | | | | | | | |
| | 0 | 0.00 | 1 | 2 | 0 | 0.00 | 4 | 10.00 |
| Yes | 0 | 0.00 | 0 | 0.00 | | 0.0 | D | 0.00 |
| No | 4 | 100.00 | 4 | 80.00 | | 70 | 9 | 90.00 |
| PU Heel L | | | | | | | | |
| Yes | 0 | | | 0.00 | 0 | 0. | Q | 0.00 |
| No | 4 | 100 | 5 | | 7 | 100.00 | | 100.00 |
| PU Troch R | | | | | | | | |
| Yes | 0 | 0.00 | | | 0 | 0.00 | 0 | 0.00 |
| N | 4 | 100.00 | | 100.00 | 1 | 100.00 | 10 | 100.00 |
| Troch L | | | 1 | | | | | |
| Yes | 0 | | 0 | .00 | 0 | 0.00 | 0 | 0.00 |
| No | | 100. | 5 | 0.00 | 1 | 100.00 | 10 | 100.00 |

Table 3. Pressure Ulcer and Randomised Arm - stratified by patient characteristics

| | | Randomised arm | | | | | |
|---|---|---|---|---|---|---|---|
| | | Treatment | | Standard of<br>Care | | 7 | Γotal |
| | | N | % | N | % | N | % |
| All | Pressure ulcer | | | | | | |
| | Yes | 2 | 22.2 | 0 | 0.0 | 2 | 20.0 |
| | No | 7 | 77.8 | 1 | 100.0 | 8 | 80.0 |
| Site | Pressure ulcer | | | | | | |
| AZ Groeninge | Yes | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | No | | 00.0 | 1 | 100.0 | 4 | 100.0 |
| UZ Brussel | Yes | 0 | | 0 | 0 | 0 | 0.0 |
| | No | 1 | 1 | 0 | 0 | 1 | 100.0 |
| Aalst | Ye | 1 | d | 0 | 0 | 1 | 50.0 |
| | No | 1 | 50.0 | 0 | 0 | 1 | 50.0 |
| AZ Zottegem | Yes | | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | | 100.0 | 0 | 0 | 1 | 100.0 |
| UZ Leuven | Yes | | 100.0 | 0 | 0 | 1 | 100.0 |
| | | 0 | | 0 | 0 | 0 | 0.0 |
| OLV Waregem | Yes | | 0.0 | 0 | 0 | 0 | 0.0 |
| | | | 100.0 | 0 | 0 | 1 | 100.0 |
| A | ressure ulcer | | | | | | |
| <60 | (es | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| 60-69 | S | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| 70-79 | Yes | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 2 | 100.0 | 0 | 0 | 2 | 100.0 |
| >=80 | Yes | 2 | 40.0 | 0 | 0.0 | 2 | 33.3 |
| | No | 3 | 60.0 | 1 | 100.0 | 4 | 66.7 |
| Gender type | Pressure ulcer | | | | | | |
| Female | Yes | 2 | 25.0 | 0 | 0.0 | 2 | 22.2 |
| | No | 6 | 75.0 | 1 | 100.0 | 7 | 77.8 |
| Male | Yes | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 1 | 100.0 | 0 | 0 | 1 | 100.0 |



Table 3. Pressure Ulcer and Randomised Arm - stratified by patient characteristics

| | | Randomised arm | | | | | |
|---|---|---|---|---|---|---|---|
| | | Trea | tment | Standard of<br>Care | | Т | otal |
| | | N | % | N | % | N | % |
| Ward type on which patient is staying (corrected) | Pressure ulcer | | | | | | |
| ICU | Yes | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| Non-ICU | Yes | 2 | 25.0 | 0 | 0.0 | 2 | 22.2 |
| | No | 6 | 75.0 | 1 | 100.0 | 7 | 77.8 |



| | | Randomised arm | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | evyn<br>ife® | Mepilex Standard Border® Care | | | T | otal | |
| | | N | % | N | % | N | % | N | % |
| All | Pressure ulcer | | | | | | | | |
| | Yes | 2 | 50.0 | 0 | 0.0 | 0 | 0.0 | 2 | 20.0 |
| | No | 2 | 50.0 | 5 | 100.0 | 1 | 100.0 | 8 | 80.0 |
| Site | Pressure ulcer | | | | | | | | |
| AZ Groeninge | Yes | 0 | 0 | 0 | 0.0 | 0 | 0.0 | 0 | 0.0 |
| | No | 0 | 0 | 3 | 100.0 | 1 | 100.0 | 4 | 100.0 |
| UZ Brussel | Yes | 0 | 0.0 | 0 | 0 | 0 | 0 | 0 | 0.0 |
| | No | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 100.0 |
| Aalst | Yes | | 50. | Q | 0 | 0 | 0 | 1 | 50.0 |
| | No | 1 | 50.0 | | 0 | 0 | 0 | 1 | 50.0 |
| AZ Zottegem | Yes | 0 | 0 | | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 0 | | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| UZ Leuven | Yes | | 0.0 | 0 | 0 | 0 | 0 | 1 | 100.0 |
| | No | | 0.0 | 0 | 0 | 0 | 0 | 0 | 0.0 |
| OLV Waregem | | 0 | | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 0 | 0 | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| Age (years) | Pressure | | | | | | | | |
| <60 | es | 0 | 0 | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | | 0 | 0 | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| 60-69 | | 0 | 0 | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 0 | 0 | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| 70-79 | Yes | 0 | 0 | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 0 | 0 | 2 | 100.0 | 0 | 0 | 2 | 100.0 |
| >=80 | Yes | 2 | 50.0 | 0 | 0.0 | 0 | 0.0 | 2 | 33.3 |
| | No | 2 | 50.0 | 1 | 100.0 | 1 | 100.0 | 4 | 66.7 |
| Gender type | Pressure ulcer | | | | | | | | |
| Female | Yes | 2 | 50.0 | 0 | 0.0 | 0 | 0.0 | 2 | 22.2 |
| | No | 2 | 50.0 | 4 | 100.0 | 1 | 100.0 | 7 | 77.8 |
| Male | Yes | 0 | 0 | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 0 | 0 | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| Ward type on which patient is staying (corrected) | Pressure ulcer | | | | | | | | |
| ICU | Yes | 0 | 0 | 0 | 0.0 | 0 | 0 | 0 | 0.0 |
| | No | 0 | 0 | 1 | 100.0 | 0 | 0 | 1 | 100.0 |
| Non-ICU | Yes | 2 | 50.0 | 0 | 0.0 | 0 | 0.0 | 2 | 22.2 |
| | No | 2 | 50.0 | 4 | 100.0 | 1 | 100.0 | 7 | 77.8 |



# APPENDIX 4. TEMPLATE TABLES RESULTS (3) HEALTH ECONOMIC OUTCOMES

| | | Randomised arm | | | |
|---|---|---|---|---|---|
| | | Allevyn<br>Life® | Mepilex<br>Border® | Standard of Care | All |
| Dressing applied - All | N | 4 | 5 | 1 | 10 |
| | Mean | 16.50 | 12.40 | 0.00 | 12.80 |
| | Std | 9.47 | 6.11 | 0 | 8.42 |
| | Min | 9.00 | 5.00 | 0.00 | 0.00 |
| | Q1 | 10.00 | 00 | 2.00 | 9.00 |
| | Median | 13.5 | 12.00 | 00 | 11.50 |
| | Q3 | | 12.00 | 00 | 16.00 |
| | Max | 34 | 22.00 | 0.00 | 30.00 |
| | NMiss | 0 | O | 0 | 0 |
| Dressing applied - Sacrum | N | 4 | | 1 | 10 |
| | | 4.00 | 3.0 | 0.00 | 3.10 |
| | Std | | 2.83 | 0 | 2.28 |
| | in | 3 | | 0.00 | 0.00 |
| | | .50 | 2.6 | 0.00 | 2.00 |
| | M. | 4.00 | 2.00 | 0.00 | 2.50 |
| | Q3 | 4.50 | 2.00 | 0.00 | 4.00 |
| | Max | 5.00 | 8.00 | 0.00 | 8.00 |
| | Miss | 0 | 0 | 0 | 0 |
| Di ned - Heel R | Ĭ | 4 | 5 | 1 | 10 |
| | ean | 4.75 | 1.80 | 0.00 | 2.80 |
| | Std | 4.57 | 1.48 | 0 | 3.33 |
| | Min | 0.00 | 0.00 | 0.00 | 0.00 |
| | Q1 | 1.00 | 1.00 | 0.00 | 0.00 |
| | Median | 4.50 | 2.00 | 0.00 | 2.00 |
| | Q3 | 8.50 | 2.00 | 0.00 | 4.00 |
| | Max | 10.00 | 4.00 | 0.00 | 10.00 |
| | NMiss | 0 | 0 | 0 | 0 |

| | | R | | | |
|---|---|---|---|---|---|
| | | Allevyn<br>Life® | Mepilex<br>Border® | Standard of Care | All |
| Dressing applied - Heel L | N | 4 | 5 | 1 | 10 |
| | Mean | 4.25 | 2.20 | 0.00 | 2.80 |
| | Std | 4.03 | 0.84 | 0 | 2.78 |
| | Min | 1.00 | 1.00 | 0.00 | 0.00 |
| | Q1 | 1.50 | 2.00 | 0.00 | 1.00 |
| | Median | 3.00 | 2.00 | 0.00 | 2.00 |
| | Q3 | 7.00 | 3.00 | 0.00 | 3.00 |
| | Max | 10.00 | 3.0 | 0.00 | 10.00 |
| | NMiss | 0 | U | 0 | 0 |
| Dressing applied - Troch R | N | A | 5 | | 10 |
| | Mean | | 2.80 | .00 | 2.00 |
| | Std | 0. | 1.48 | 0 | 1.41 |
| | Min | 1.00 | | 0.00 | 0.00 |
| | Q1 | 1.00 | | 0.00 | 1.00 |
| | | 1.50 | 3.00 | 0.00 | 2.00 |
| | <b>Q</b> 3 | | 3.00 | 0.00 | 3.00 |
| <b>\</b> | ιx | | | 0.00 | 5.00 |
| | ss | 0 | 0 | 0 | 0 |
| Dress' Troch L | N | 4 | 5 | 1 | 10 |
| | Mea | 2.00 | 2.60 | 0.00 | 2.10 |
| | Std | 1.83 | 2.70 | 0 | 2.23 |
| | in | 0.00 | 0.00 | 0.00 | 0.00 |
| | | 0.50 | 1.00 | 0.00 | 0.00 |
| | ledian | 2.00 | 2.00 | 0.00 | 1.50 |
| | Q3 | 3.50 | 3.00 | 0.00 | 3.00 |
| | Max | 4.00 | 7.00 | 0.00 | 7.00 |
| | NMiss | 0 | 0 | 0 | 0 |

# APPENDIX 5. TEMPLATE TABLES RESULTS (4) SAFETY OUTCOMES

| | | Intervention group | | | | | |
|---|---|---|---|---|---|---|---|
| | | Allevyn<br>Life® | | Mepilex<br>Border® | | Total | |
| | | N | % | N | % | N | % |
| All | Adverse devise effect | | | | | | |
| | Yes | | | | | | |
| | No | | | | | | |
| Site | Adverse devise effect | | | | | | |
| UZ Gent | Yes | | | | | | |
| | No | | | | | | |
| AZ Groeninge | Yes | | | | | | |
| | No | | | | | | |
| UZ Brussel | Yes | | | | | | |
| | No | | abla | | | | |
| Aalst | Yes | | | | | | |
| | No | | | | | | |
| AZ Zottegem | Yes | | | | | | |
| | No | | | | | | |
| UZ Leuven | Yes | | | | | | |
| | No | | | | | | |
| Magniddelares | Yes | | | | | | |
| OL Grego | ıes | | | | | | |
| | No | | | | | | |

| Ye | evise deficiency<br>es | Alle<br>Li<br>N | evyn<br>fe®<br>% | Mer<br>Bor | oilex<br>der®<br>% | To<br>N | otal<br>% |
|---|---|---|---|---|---|---|---|
| Site De UZ Gent Ye | | N | % | N | % | N | % |
| Site De UZ Gent Ye | | | | | | | |
| Site De UZ Gent Ye | es | | | | | | |
| Site De UZ Gent Ye | | 65 | 12.0 | 32 | 5.9 | 97 | 8.9 |
| UZ Gent Ye | 0 | 478 | 88.0 | 513 | 94.1 | 991 | 91.1 |
| | evise deficiency | | | | | | |
| NI. | es | | | | <u> </u> | | |
| NO | 0 | | | | | | |
| AZ Groeninge Ye | es | | 47 | | | | |
| No | 0 | | | | | | |
| UZ Brussel Ye | es | | | | | | |
| No | 0 | | | | | | |
| Aalst Ye | es | | | | | | |
| No | | | | | | | |
| AZ Zottegem Ye | es | | | | | | |
| No | 0 | | | | | | |
| UZ Leuven Ye | es | | | | | | |
| No | 0 | | | | | | |
| Mari Ye | es | | | | | | |
| No | 0 | | | | | | |
| V Waregem | | | | | | | |
| No | | | | | | | |

